CLINICAL TRIAL: NCT02312999
Title: Phase IV, Multicentric, Prospective, Controlled, Randomized, Double Blind Study Comparing a Crystalloid to a Colloid Used in the Perioperatory Hemodynamic Optimisation With a 'Closed Loop' Automatic Filling System, on the Post-surgery Morbidity in Major Abdominal Surgery.
Brief Title: Crystalloids or Colloids for Goal-directed Fluid Therapy With Closed-loop Assistance in Major Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Philippe VAN DER LINDEN, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUB-fluides
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Surgery
Keywords: laparotomy; plasma-Lyte; volulyte; close loop; abdominal surgery
MeSH Terms: interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volulyte (Experimental): A baseline crystalloid infusion (plasmalyte®) will be set by the attending physician at 3 cc/kg/hr (standard patient care) for each of the randomized groups. The patient will receive fluid management via a closed loop (automated) system that will use an infusion pump (Q-Core) and a controller (a computer run index and algorithm developed by Sironis) to standardize the way fluids are administered intra-operatively and eliminate variation between clinical providers. The liquid perfused will be bolus amounts of volulyte.
  Interventions: Drug: Volulyte
- Plasma-Lyte (Active Comparator): A baseline crystalloid infusion (plasmalyte®) will be set by the attending physician at 3 cc/kg/hr (standard patient care) for each of the randomized groups. The patient will receive fluid management via a closed loop (automated) system that will use an infusion pump (Q-Core) and a controller (a computer run index and algorithm developed by Sironis) to standardize the way fluids are administered intra-operatively and eliminate variation between clinical providers. The liquid perfused will be bolus amounts of plasma-lyte.
  Interventions: Drug: Plasmalyte

INTERVENTIONS:
Drug: Plasmalyte
  Arms: Plasma-Lyte
Drug: Volulyte
  Arms: Volulyte

SUMMARY:
Study goal: This study will examine whether there is a significant difference in postoperative outcomes between GDFT using a colloid solution versus a crystalloid solution.

Hypothesis: Perioperative fluid optimization through the use of a closed-loop assistance with a balanced starch solution (volulyte®) will be associated with a decrease in postoperative complications compared to the same approach using a balanced crystalloid solution (Plasmalyte®).

Objective: To establish which kind of intravenous fluid used for goal directed therapy with closed-loop assistance will reduce the number of postoperative complications (evaluation made by the POMS score).

DETAILED DESCRIPTION:
Controversy still persists regarding the type of fluid to use in the operating room to avoid hypovolemia and any circulatory insufficiency. While crystalloids and colloid solutions are frequently used to optimize intravascular volume during surgery, crystalloid solutions require more volume for hemodynamic optimization which may result in higher volumes of fluid administration and potentially side effects. Compared with crystalloids, colloids have the advantages of remaining in the intravascular space longer, achieving faster circulatory stabilization, maintaining colloid osmotic pressure and increasing micro perfusion. However, colloids are more expensive and may have various side effects.

In addition to the effect of crystalloids and colloids on the patient, the amount of each fluid administered is also under debate. Goal-directed fluid therapy (GDFT) strategies based on cardiac output (CO) optimization have been shown to benefit moderate- to high-risk surgery patients and have recently been recommended by professional societies in the UK, in France, and in Europe. However, despite the growing evidence, these strategies are often not implemented in current practice. One of the reasons for this lack of implementation is that GDFT strategies, like any other complex clinical protocol, require significant provider attention and vigilance for consistent implementation and it is well known that even under study conditions protocol compliance rates are often not greater than 50% In another hand, one of the chief complicating factors in fluid administration studies is variation in provider administration practices, even when attempting to follow a protocol. Previous studies have used closed-loop (automated) systems to deliver fluid by a standardized protocol, removing variation between providers as one of the confounders of the study. Dr. Cannesson and Rinehart (UC Irvine, California, USA) have recently developed and used a closed-loop system for the provision of GDFT in clinical studies at UC Irvine and La Pitie hospital in France. The closed-loop system is beneficial because it involves the standardization of fluid management and all patients are treated equivalently. This system will thus provide consistent GDFT for all cases in the protocol and remove inter-provider variability as a confounder between groups.

Study goal: This study will examine whether there is a significant difference in postoperative outcomes between GDFT using a colloid solution versus a crystalloid solution.

Hypothesis: Perioperative fluid optimization through the use of a closed-loop assistance with a balanced starch solution (volulyte®) will be associated with a decrease in postoperative complications compared to the same approach using a balanced crystalloid solution (Plasmalyte®).

Objective: To establish which kind of intravenous fluid used for goal directed therapy with closed-loop assistance will reduce the number of postoperative complications (evaluation made by the POMS score).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over the age of 18) undergoing elective major abdominal surgery that is expected to take longer than 3 hours and requiring a general anesthesia and a minimally invasive cardiac output monitoring (Vigileo/Flotrac)
* Patients who provide written informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients not undergoing surgery, requiring anesthesia, or cardiac output monitoring
* Patients with arrhythmia and/or atrial fibrillation
* Patients who are allergic to HES
* Patients with renal insufficiency (serum creatinine of >2 mg/ml) or hepatic dysfunction (liver enzymes >1.5)
* Patients who has coagulation disorders (please define: values higher than 1.5x normal values
* Patients without the capacity to give written informed consent or refusal of consent
* Patients included in another protocol within a period of 3 months or Participating in another randomised trial
* Pregnancy at time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
POMS score | 48 hours
  Difference between the 2 groups in postoperative morbidity identified with the Post-Operative Morbidity Survey (POMS score) on postoperative days 2.

SECONDARY OUTCOMES:
Mortality rate | 30 days
  Difference in 30-day post-operative mortality between the 2 groups
Length of hospitalisation | every day up to 90 days after hospitalisation
  Difference in duration of hospital length of stay as well as ICU length of stay.
Quantity of fluid administered during surgery | 24 hours
  Fluid balance during surgery
Transfusion rate | 8 days
  Differences of transfusion rate between the two groups, in ml
Hypotension incidence | 8 days
  Incidence of hypotension (defined as total case time spent with 20% drop from baseline preoperative blood pressure).
Need of vasopressors | 24 hours
  Difference in the need and quantity of vasopressors between the two groups
Mean case cardiac index (L /BSA) | 24 hours
  Mean case cardiac index (L /BSA), Mean case cardiac stroke volume index (mL/ BSA).
Whodas scale | 6 months after surgery
  Enrolled patients will be contacted by phone and their quality of life assessed by the Whodas scale
Whodas scale | 1 year after surgery
  Enrolled patients will be contacted by phone and their quality of life assessed by the Whodas scale
Pruritus apparition | 6 months after surgery
  Enrolled patients will be contacted by phone 6 months after surgery and any pruritus apparition will be recorded
Pruritus apparition | 1 year after surgery
  Enrolled patients will be contacted by phone 1 year after surgery and any pruritus apparition will be recorded
Renal function - urea level | 6 months after surgery
  Urea levels. Measured in a blood sample taken according to the standard of care outpatient post-operative follow appointments.
Renal function - urea level | 1 year after surgery
  Urea levels. Measured in a blood sample taken according to the standard of care outpatient post-operative follow appointments.
Renal function - creatinine level | 6 months after surgery
  Creatinine levels. Measured in a blood sample taken according to the standard of care outpatient post-operative follow appointments.
Renal function - creatinine level | 1 year after surgery
  Creatinine levels. Measured in a blood sample taken according to the standard of care outpatient post-operative follow appointments.
Renal function - Estimated glomerular filtration rate (eGFR) | 6 months after surgery
  Creatinine levels. Measured in a blood sample taken according to the standard of care outpatient post-operative follow appointments.
Renal function - Estimated glomerular filtration rate (eGFR) | 1 year after surgery
  Creatinine levels. Measured in a blood sample taken according to the standard of care outpatient post-operative follow appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Delaporte, MD, Principal Investigator — CHU Brugmann; Alexandre Joosten, MD, Principal Investigator — Erasme; Philippe Van der Linden, MD, Pr, Principal Investigator — CHU Brugmann; Brigitte Ickx, Md, Pr, Principal Investigator — Erasme
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - Erasme, Brussels

REFERENCES:
- [Background] Feldheiser A, Pavlova V, Bonomo T, Jones A, Fotopoulou C, Sehouli J, Wernecke KD, Spies C. Balanced crystalloid compared with balanced colloid solution using a goal-directed haemodynamic algorithm. Br J Anaesth. 2013 Feb;110(2):231-40. doi: 10.1093/bja/aes377. Epub 2012 Oct 30. PMID 23112214
- [Background] Silva JM Jr, de Oliveira AM, Nogueira FA, Vianna PM, Pereira Filho MC, Dias LF, Maia VP, Neucamp Cde S, Amendola CP, Carmona MJ, Malbouisson LM. The effect of excess fluid balance on the mortality rate of surgical patients: a multicenter prospective study. Crit Care. 2013 Dec 10;17(6):R288. doi: 10.1186/cc13151. PMID 24326085
- [Background] Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, Madsen KR, Moller MH, Elkjaer JM, Poulsen LM, Bendtsen A, Winding R, Steensen M, Berezowicz P, Soe-Jensen P, Bestle M, Strand K, Wiis J, White JO, Thornberg KJ, Quist L, Nielsen J, Andersen LH, Holst LB, Thormar K, Kjaeldgaard AL, Fabritius ML, Mondrup F, Pott FC, Moller TP, Winkel P, Wetterslev J; 6S Trial Group; Scandinavian Critical Care Trials Group. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. N Engl J Med. 2012 Jul 12;367(2):124-34. doi: 10.1056/NEJMoa1204242. Epub 2012 Jun 27. PMID 22738085
- [Background] Cannesson M. Arterial pressure variation and goal-directed fluid therapy. J Cardiothorac Vasc Anesth. 2010 Jun;24(3):487-97. doi: 10.1053/j.jvca.2009.10.008. No abstract available. PMID 20022261
- [Background] Ramsingh DS, Sanghvi C, Gamboa J, Cannesson M, Applegate RL 2nd. Outcome impact of goal directed fluid therapy during high risk abdominal surgery in low to moderate risk patients: a randomized controlled trial. J Clin Monit Comput. 2013 Jun;27(3):249-57. doi: 10.1007/s10877-012-9422-5. Epub 2012 Dec 22. PMID 23264068
- [Background] Pearse RM, Harrison DA, MacDonald N, Gillies MA, Blunt M, Ackland G, Grocott MP, Ahern A, Griggs K, Scott R, Hinds C, Rowan K; OPTIMISE Study Group. Effect of a perioperative, cardiac output-guided hemodynamic therapy algorithm on outcomes following major gastrointestinal surgery: a randomized clinical trial and systematic review. JAMA. 2014 Jun 4;311(21):2181-90. doi: 10.1001/jama.2014.5305. PMID 24842135